CLINICAL TRIAL: NCT04497337
Title: The Superficial Lesions in the Peri-auricular Region; Retrospective Study
Brief Title: The Superficial Lesions in the Peri-auricular Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed Elrabie Ahmed (Other)
Responsible Party: Sponsor-Investigator, Mohammed Elrabie Ahmed, Clinical Professor of Otolarygology head and neck surgery, Sohag University
Organization: Sohag University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18630159
Record Dates: First submitted 2020-07-27; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Superficial Cyst or Mass and Sinus on and Around the Ear
MeSH Terms: conditions — Arachnodactyly

STUDY DESIGN:
Intervention Model Description: Data included in this descriptive retrospective study were collected from records of 70 patients with superficial lesions around the auricle, i.e., periauricular (preauricular, auricular, and postauricular) during the period extending between 2017 and 2019, who were primarily diagnosed and operated
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Complete excision to superficial lesions around the ear — Complete excision of these lesions and histopathology

SUMMARY:
Superficial lesions on and around the ear are uncommon with many differential diagnoses and different characteristic histopathologic features. The purpose of this study was to describe a series of peri-auricular superficial lesions and characterize the distinctive types of these lesions.

DETAILED DESCRIPTION:
Data included in this descriptive retrospective study were collected from records of 70 patients with superficial lesions around the auricle, i.e., periauricular (preauricular, auricular, and postauricular) during the period extending between 2017 and 2019, who were primarily diagnosed and operated. Data were retrieved, reviewed, and analyzed. The primary analysis outcome measures were patient history (age, gender, complaint, medical advice clinic, and associated medical diseases), lesions examination (site, laterality, clinical presentation, and the number of lesions). Also, the needed investigations for diagnosis, type of intervention, postoperative patient satisfaction were evaluated. Evaluation of the patients' follow up was done.

ELIGIBILITY:
Inclusion Criteria:

* Patients with superficial lesions around the auricle, i.e., periauricular (preauricular, auricular, and postauricular) operated during the period extending between 2017 and 2019
* Available full demographic, clinical and histopathological data

Exclusion Criteria:

* deep lesions involving parotid or parapharyngeal space
* Missed demographic, clinical and histopathological data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-05-16 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
clinical and Histopathlogical types of superficial lesion around the ear | Cases operated between in the previous 3 years from 2017 and 2019

CONTACTS AND LOCATIONS:
Overall Officials: Sohag University hospital, Study Director — Nasr City, Eastern Avenue, University Street, Sohag, Egypt
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided